CLINICAL TRIAL: NCT04959188
Title: Needs Assessment for Individuals and Families Affected by Dyskeratosis Congenita (DC) and Related Telomere Biology Disorders (TBD)
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000502; 000502-C
Record Dates: First submitted 2021-07-10; First posted 2021-07-13 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12-09

CONDITIONS: Dyskeratosis Congenita; Telomere Biology Disorders
Keywords: Online Survey; Qualitative Interviews; germline variants; Bone Marrow Failure; Natural History
MeSH Terms: conditions — Dyskeratosis Congenita; Bone Marrow Failure Disorders

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Bereaved family caregivers: Bereaved family caregivers (parents or spouses/partners) of individuals who died from complications associated with dyskeratosis congenita or a related telomere biology disorder.
- Caregivers: Family and/or caregivers of individuals with dyskeratosis congenita or a related telomere biology disorder.
- Patients: Individuals with dyskeratosis congenita or a related telomere biology disorder.

SUMMARY:
Background:

DC and related TBDs are a group of illnesses caused by variants in genes that regulate telomeres. These illnesses can cause problems with the skin and mucous membranes. They can also cause ophthalmic, dental, immunologic, and other abnormalities. Researchers want to learn more about these illnesses and the people who have them.

Objective:

To learn about the informational, pragmatic, and psychosocial challenges and unmet needs of individuals and families affected by DC and related TBDs.

Eligibility:

People aged 18 years and older who have DC or related TBD or who are, or have been, a caregiver to someone with DC or related TBD.

Design:

This study has 2 parts: a survey and a telephone interview. Participants may choose to take part in one or both parts.

Participants may complete an online survey. They will select which group most applies to them: person with DC/TBD; parent/caregiver to a person with DC/TBD; or bereaved parent/caregiver of a person who had DC/TBD. The survey will be based on the group they choose. They will answer 20-30 questions. The survey will take 10-20 minutes to complete.

Participants may take part in a phone interview. It will take 50-70 minutes to complete. They will give their name, email address, and phone number to schedule the interview. The interview will be audio recorded and transcribed. Personal identifiers will be removed.

DETAILED DESCRIPTION:
Study Description:

This study is exploratory and aims to conduct a needs assessment for individuals and families living with DC and related TBDs. The study has two parts. For the first part of the study, participants will complete an online survey. The second part of the study involves participating in an interview via telephone. Interviews will address important questions in greater depth. Individuals have the option to participate in one or both parts of the study.

Objective:

Using online survey methodology and qualitative interviews, the purpose of this concurrent mixed methods study is to conduct a needs assessment about the informational, pragmatic, and psychosocial challenges and unmet needs of individuals and families affected by DC and related TBDs.

Endpoint:

This is an exploratory study; therefore, we are not generating a priori hypotheses. Statistical analysis will be limited to calculating descriptive statistics (frequencies, percentages, chi-square statistics) and statistical analyses that do not require a large number of observations (Pearson's r, ANOVA).

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet the following criteria:

* Ability for the participant to speak, read, and/or write in English to understand and sign the informed consent and complete the online survey, interview, or both.
* Participants must have a diagnosis of DC or related TBD or be, or have been, a caregiver to an individual with a diagnosis of DC or related TBD.
* Participants must be 18 years of age or older.
* Participants must have Internet access to participate in the online survey and a telephone to participate in the interview.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

-Individuals who do not meet eligibility criteria listed above. No other exclusionary criteria apply.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals and families living with DC or a related TBD from relevant patient advocacy groups or referred by colleagues or professional groups.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2021-09-09 (Actual); Primary Completion 2023-07-05 (Actual); Study Completion 2023-07-05 (Actual)

PRIMARY OUTCOMES:
Needs Assessment | Will be ongoing while the study is open
  Brief online survey consisting of questions that have been modified from the Needs Assessment of Family Caregivers-Cancer (NAFC-C) which has been validated in caregiver and bereaved populations.

SECONDARY OUTCOMES:
Needs assessment | Will be ongoing while the study is open
  Semi-structured interview guide; 60 to 90 minute telephone interviews to assess the needs of patients and their families and caregivers

CONTACTS AND LOCATIONS:
Overall Officials: Sharon A Savage, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Niewisch MR, Savage SA. An update on the biology and management of dyskeratosis congenita and related telomere biology disorders. Expert Rev Hematol. 2019 Dec;12(12):1037-1052. doi: 10.1080/17474086.2019.1662720. Epub 2019 Sep 10. PMID 31478401
- [Background] Hamilton JG, Hutson SP, Frohnmayer AE, Han PK, Peters JA, Carr AG, Alter BP. Genetic Information-Seeking Behaviors and Knowledge among Family Members and Patients with Inherited Bone Marrow Failure Syndromes. J Genet Couns. 2015 Oct;24(5):760-70. doi: 10.1007/s10897-014-9807-3. Epub 2014 Dec 27. PMID 25540896
- [Background] Hutson SP, Han PK, Hamilton JG, Rife SC, Al-Rahawan MM, Moser RP, Duty SP, Anand S, Alter BP. The use of haematopoietic stem cell transplantation in Fanconi anaemia patients: a survey of decision making among families in the US and Canada. Health Expect. 2015 Oct;18(5):929-41. doi: 10.1111/hex.12066. Epub 2013 Apr 29. PMID 23621292